CLINICAL TRIAL: NCT05517031
Title: Unmet Needs of Axial Spondyloarthrits in Egyptian Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Toqa Mahfouz Mohamed Ahmed, Resident doctor at rheumatology and rehabilitation department faculty of medicine Sohag university, Sohag University
Other Study IDs: Soh-Med-22-08-04
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ASDAS score , VAS score, BASFI score , Katz ADL index — Scores that done on patient to fullfill criteria of diagnosis , and measure affection of disease on patients and their daily living activity

SUMMARY:
During the past decade, the well-known disease called Ankylosing Spondylitis has come to be considered as a subset of the broader entity referred as axial spondyloarthritis (axSpA), which also includes non-radiographic axSpA. The need of this new classification was aimed to improve the sensitivity for an early diagnosis, to reduce diagnostic delay, and to allow an early treatment. Although there is improvement in the recognition, the management of patients, and the treatment strategies of axSpA, unmet needs persist , there is still a substantial gap of 5-8 years between the onset of symptoms and the diagnosis of axSpA.

. This study is intended to enhance awareness and understanding of Axial Spondyloarthritis and to identify and discuss the current unmet needs in axSpA .

Multiple defects are still unfullfilled for axial SpA patients those defects include delayed diagnosis specially for female, failure to acheive treatment target, pain, impaired quality of life and associated comorbidities.

Up to the best of our knowledge this is the first study to highlight unmet needs for axial Spondyloarthritis patients in Egypt in general and in upper Egypt in particular .

ELIGIBILITY:
Inclusion Criteria

* Patients fulfill the Assessment in Spondyloarthrits International Society (ASAS) classification criteria for Axial Spondyloarthritis .
* Age above 16 years old.
* Patient cooperative and can answer questions .

Exclusion Criteria:

* Other rheumatologic or collagen diseases .
* Age below 16 years and above 60 years.
* Uncooperative patients .

Ages: 16 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients fulfill the Assessment in Spondyloarthrits International Society (ASAS) classification criteria for Axial Spondyloarthritis With comorbidities as diabetes , hypertension , pregnancy , renal impairment or smoking
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
(ASDAS score ) The Ankylosing Spondylitis Disease Activity score | 3 months
  an index to assess disease activity in Ankylosing Spondylitis (AS).
(VAS score ) Visual Analogue Score | 3 months
  A psychometric response scale for parameters that range across a continuum of values, such as pain. The VAS pain scale ranges from "no pain" to "worst pain," and patients mark a line to indicate how they are feeling.
(BASFI score ) Bath Ankylosing Spondylitis Functional Index | 3 months
  The BASFI consists of 10 questions, answered on a VAS. The final score is the average of the questions, ranging from 0 (no limitation) to 10 (maximal limitation in function).
Katz Activity Daily Living | 3 months
  The Katz Activities of Daily Living (ADL) scale is a widely used graded instrument that assesses six primary and psychosocial functions: bathing, dressing, going to toilet, transferring, feeding, and continence.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Landewe R, Braun J, Deodhar A, Dougados M, Maksymowych WP, Mease PJ, Reveille JD, Rudwaleit M, van der Heijde D, Stach C, Hoepken B, Fichtner A, Coteur G, de Longueville M, Sieper J. Efficacy of certolizumab pegol on signs and symptoms of axial spondyloarthritis including ankylosing spondylitis: 24-week results of a double-blind randomised placebo-controlled Phase 3 study. Ann Rheum Dis. 2014 Jan;73(1):39-47. doi: 10.1136/annrheumdis-2013-204231. Epub 2013 Sep 6. PMID 24013647
- [Background] Kiltz U, Heldmann F, Baraliakos X, Braun J. Treatment of ankylosing spondylitis in patients refractory to TNF-inhibition: are there alternatives? Curr Opin Rheumatol. 2012 May;24(3):252-60. doi: 10.1097/BOR.0b013e3283524b82. PMID 22450391
- [Background] Hamilton L, Barkham N, Bhalla A, Brittain R, Cook D, Jones G, Mackay K, Marshall D, Marzo-Ortega H, Murphy D, Riddell C, Sengupta R, Siebert S, Van Rossen L, Gaffney K; BSR and BHPR Standards, Guidelines and Audit Working Group. BSR and BHPR guideline for the treatment of axial spondyloarthritis (including ankylosing spondylitis) with biologics. Rheumatology (Oxford). 2017 Feb;56(2):313-316. doi: 10.1093/rheumatology/kew223. Epub 2016 Aug 24. No abstract available. PMID 27558584
- [Background] Rudwaleit M, van der Heijde D, Landewe R, Listing J, Akkoc N, Brandt J, Braun J, Chou CT, Collantes-Estevez E, Dougados M, Huang F, Gu J, Khan MA, Kirazli Y, Maksymowych WP, Mielants H, Sorensen IJ, Ozgocmen S, Roussou E, Valle-Onate R, Weber U, Wei J, Sieper J. The development of Assessment of SpondyloArthritis international Society classification criteria for axial spondyloarthritis (part II): validation and final selection. Ann Rheum Dis. 2009 Jun;68(6):777-83. doi: 10.1136/ard.2009.108233. Epub 2009 Mar 17. PMID 19297344